CLINICAL TRIAL: NCT01861925
Title: Lenstar LS 900 Topography
Brief Title: Study of Clinical Performance of Corneal Topography Measurement Using an Optical Biometer
Status: Completed | Type: Observational
Sponsor: Haag-Streit AG (Industry)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: HS-LS900-TOPO-01
Record Dates: First submitted 2013-05-21; First posted 2013-05-24 (Estimated); Results first posted 2014-06-05 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-05

CONDITIONS: Corneal Topography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Normal eye: Astigmatism smaller than 1.5 diopters
- Large regular astigmatism: Astigmatism of > 1.5 diopters, regular astigmatism.
- Large irregular astigmatism: Astigmatism of > 1.5 diopters, irregular astigmatism.

SUMMARY:
The purpose of this study is to quantify in-vivo repeatability of a new corneal topography measurement mode of an optical biometer, and the clinical performance of measurement in comparison to reference devices.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older

Exclusion Criteria:

* No corneal transplants
* No corneal scar(s)
* No acute infections of the eye
* No weak fixation
* No suspected lack of compliance
* No vulnerable population

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers recruited at University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Frueh, Prof. Fr., Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- University Hospital Inselspital, Bern, Switzerland

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Normal Eye | Large Regular Astigmatism | Large Irregular Astigmatism
Started | 34 | 8 | 8
Completed | 34 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Eye | Large Regular Astigmatism | Large Irregular Astigmatism | Total
Number analyzed (Participants) | 34 | 8 | 8 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (9.8) | 36.4 (9.0) | 32.7 (8.2) | 37.4 (9.5)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 34 | 8 | 8 | 50
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 2 | 0 | 15
  Male | 21 | 6 | 8 | 35
Region of Enrollment [Number; unit: participants]
  Switzerland | 34 | 8 | 8 | 50

OUTCOME MEASURES:

1. Primary Outcome: In-vivo Repeatability of Corneal Topography Measurements With Lenstar LS 900 Topography: Sample Mean of Differences of Mean Power and Sample Mean of Std. Dev of Local Power Differences Between Two Consecutive Measurements
Description: Corneal topography is a measurement of the shape of the anterior cornea. The shape of a cornea can be fully quantified by providing a map of local power. "Diopter" is the unit of refractive power of a lens. In case of the cornea, the power K [diopter] is related to the radius (curvature) R [mm] of the best fitting sphere by the relation K=337.5/R.
  Here, corneal topography measurements are implemented by the Placido method, i.e. by analyzing the reflection image of a ring-shaped illumination.
  According to International Standards Organization (ISO) 19980-2012, repeatability of corneal topography is assessed on the central cornea: area with diameter d<=3mm, and middle cornea: 3mm<d<=6mm.
  "power difference (2 rep. meas.)": sample mean and 95% C.I. of differences of spatial mean of corneal power between two consecutive measurements.
  "power difference 2 std.dev.": sample mean of twice the deviation of local power differences (two consecutive measurements).
Time Frame: 1 day of examination
Measure: Mean (95% Confidence Interval); unit: diopters
Arm/Group | Normal Eye | Large Regular Astigmatism | Large Irregular Astigmatism
Number analyzed (Participants) | 34 | 8 | 8
diopters
  power difference (2 rep. meas.), central cornea | -0.014 [-0.062 to 0.034] | 0.053 [-0.061 to 0.167] | -0.120 [-0.392 to 0.153]
  power difference (2 rep. meas.), middle cornea | -0.029 [-0.090 to 0.033] | 0.015 [-0.149 to 0.179] | -0.089 [-0.351 to 0.174]
  power difference (2 std.dev.), central cornea | 0.77 [NA to NA] — 95% C.I. of Std.Dev. not required by ISO 19980-2012 | 0.74 [NA to NA] — 95% C.I. of Std.Dev. not required by ISO 19980-2012 | 1.36 [NA to NA] — 95% C.I. of Std.Dev. not required by ISO 19980-2012
  power difference (2 std.dev.), middle cornea | 0.72 [NA to NA] — 95% C.I. of Std.Dev. not required by ISO 19980-2012 | 0.69 [NA to NA] — 95% C.I. of Std.Dev. not required by ISO 19980-2012 | 1.06 [NA to NA] — 95% C.I. of Std.Dev. not required by ISO 19980-2012

2. Secondary Outcome: Equivalence of Corneal Topography Measurement Between Lenstar LS 900 Topography and Atlas 9000: Sample Mean of Differences of Mean Power and Sample Mean of Std. Dev of Local Power Differences for One Measurement Per Device.
Description: For definition of corneal topography, corneal power in "diopter", areas of evaluation and methods, see outcome 1.
  This outcome measure aims at testing the equivalence of corneal topography measurement between Lenstar LS 900 Topography (Haag Streit) and Atlas 9000 (Zeiss) by analyzing differences in measurement results for the same eye between both devices.
  "power difference (2 devices)" is the sample mean and 95% C.I. of differences of spatial mean of corneal power between two devices. This value quantifies systematic differences between devices (e.g. calibration), ignoring local variations of the power measurement.
  "power difference (2 std.dev.)" is the sample mean of twice the standard deviation of local power differences between measurements with both devices. This value quantifies the spatially resolved agreement of corneal shape measurement of the two devices.
Time Frame: 1 day of examination
Measure: Mean (95% Confidence Interval); unit: diopters
Arm/Group | Normal Eye | Large Regular Astigmatism | Large Irregular Astigmatism
Number analyzed (Participants) | 34 | 8 | 8
diopters
  power difference (2 devices), central cornea | 0.044 [-0.023 to 0.110] | 0.012 [-0.039 to 0.063] | 0.160 [-0.57 to 0.889]
  power difference (2 std.dev.), central cornea | 0.79 [NA to NA] — 95% C.I. of Std.Dev. not required by ISO 19980-2012 | 0.77 [NA to NA] — 95% C.I. of Std.Dev. not required by ISO 19980-2012 | 2.49 [NA to NA] — 95% C.I. of Std.Dev. not required by ISO 19980-2012
  power difference (2 devices), middle cornea | 0.070 [-0.004 to 0.144] | 0.038 [-0.058 to 0.134] | -0.083 [-0.701 to 0.536]
  power difference (2 std.dev.), middle cornea | 0.76 [NA to NA] — 95% C.I. of Std.Dev. not required by ISO 19980-2012 | 0.72 [NA to NA] — 95% C.I. of Std.Dev. not required by ISO 19980-2012 | 1.56 [NA to NA] — 95% C.I. of Std.Dev. not required by ISO 19980-2012

3. Other Pre Specified Outcome: Equivalence of Corneal Topography Measurement Between Lenstar LS 900 Topography and Atlas 9000: Sample Mean of Std. Dev. of Local Corneal Elevation Differences for One Measurement Per Device.
Description: For definition of corneal topography, areas of evaluation and methods, see outcome 1 and 2.
  Corneal elevation refers to the distance between the measured corneal surface and the best fitting sphere, and is given in µm.
  This outcome measure aims at testing the equivalence of corneal topography measurement between Lenstar LS 900 Topography (Haag Streit) and Atlas 9000 (Zeiss) by analyzing differences in measurement results for the same eye between both devices.
  "elevation difference (2 std. dev.)" is the sample mean of twice the standard deviation of local corneal elevation differences between measurements with both devices. This value quantifies the spatially resolved agreement of corneal shape measurement of the two devices.
Time Frame: 1 day of examination
Measure: Mean (95% Confidence Interval); unit: micrometer
Arm/Group | Normal Eye | Large Regular Astigmatism | Large Irregular Astigmatism
Number analyzed (Participants) | 34 | 8 | 8
micrometer
  elevation difference (2 std. dev.), centr. cornea | 2.00 [NA to NA] — 95% C.I. of Std.Dev. not required by ISO 19980-2012 | 1.84 [NA to NA] — 95% C.I. of Std.Dev. not required by ISO 19980-2012 | 5.72 [NA to NA] — 95% C.I. of Std.Dev. not required by ISO 19980-2012
  elevation difference (2 std. dev.), middle cornea | 2.92 [NA to NA] — 95% C.I. of Std.Dev. not required by ISO 19980-2012 | 3.08 [NA to NA] — 95% C.I. of Std.Dev. not required by ISO 19980-2012 | 12.59 [NA to NA] — 95% C.I. of Std.Dev. not required by ISO 19980-2012

4. Other Pre Specified Outcome: Equivalence of Keratometry Radius Measurement Between Lenstar LS 900 Topography and Lenstar LS 900: Population Mean of Differences of Keratometry Radius Measurement Between Both Devices.
Description: Keratometry radius refers to the corneal curvature R (see primary measure outcome). In this context, the cornea is approximated by a toric surface which can be characterized by a flat meridian (radius R1) and a steep meridian (radius R2) with an angle of 90 degrees between these meridians.
  This outcome measure aims at testing the equivalence of keratometry radius measurement between Lenstar LS 900 Topography and Lenstar LS 900 (both Haag Streit) by analyzing differences in measurement results for the same eye between both devices.
  Reported are: population mean of difference and 95% confidence interval of mean difference for radius of flat meridian (R1) and radius of steep meridian (R2).
Time Frame: 1 day of examination
Measure: Mean (95% Confidence Interval); unit: micrometer
Arm/Group | Normal Eye | Large Regular Astigmatism | Large Irregular Astigmatism
Number analyzed (Participants) | 34 | 8 | 8
micrometer
  difference of flat meridian (R1) | 2.00 [-3.39 to 7.38] | -2.59 [-21.98 to 16.8] | -28.06 [-61.45 to 5.33]
  difference of steep meridian (R2) | -5.23 [-12.95 to 2.49] | -1.63 [-12.57 to 9.32] | -59.19 [-131.29 to 12.92]

5. Other Pre Specified Outcome: Equivalence of Keratometry Axis Measurement Between Lenstar LS 900 Topography and Lenstar LS 900: Population Mean of Differences of Keratometry Axis Measurement Between Both Devices.
Description: Keratometry axis refers to the axis of the flat meridian of the toric representation of the cornea. For additional information see outcome 4.
  This outcome measure aims at testing the equivalence of keratometry axis measurement between Lenstar LS 900 Topography and Lenstar LS 900 (both Haag Streit) by analyzing differences in measurement results for the same eye between both devices.
  Reported are: population mean of difference and 95% confidence interval of mean difference for axis of flat meridian.
Time Frame: 1 day of examination
Measure: Mean (95% Confidence Interval); unit: degree
Arm/Group | Normal Eye | Large Regular Astigmatism | Large Irregular Astigmatism
Number analyzed (Participants) | 34 | 8 | 8
degree | -0.13 [-1.85 to 1.59] | -0.44 [-2.02 to 1.14] | 0.25 [-3.83 to 4.34]

6. Post Hoc Outcome: Equivalence of Keratometry Axis Measurement Between Lenstar LS 900 Topography and Lenstar LS 900: Population Mean of Normalized Differences of Keratometry Axis Measurement Between Both Devices.
Description: For definition of keratometry axis see outcome measures 4 and 5.
  This outcome measure aims at testing the equivalence of keratometry axis measurement between Lenstar LS 900 Topography and Lenstar LS 900 (both Haag Streit) by analyzing differences in measurement results for the same eye between both devices.
  Reported are: population mean of normalized difference and 95% confidence interval of mean normalized difference for axis of flat meridian.
  Difference is normalized for each eye as function of astigmatism to a refractive error of 0.167 diopters (i.e. an axis difference of 1 normalized degree results in a refractive error of 0.167 diopter), to provide a measure which can be directly related to its impact on visual quality.
  Please note that for this analysis a separation in arms "normal eye" and "large regular astigmatism" is not meaningful, thus here both groups are analyzed jointly as group "regular eye"
Time Frame: 1 day of examination
Measure: Mean (95% Confidence Interval); unit: normalized degree
Groups:
- Regular Eye: Astigmatism smaller than 1.5 diopters and regular astigmatism >= 1.5 diopters (group "normal eye" and "large regular astigmatism")
Arm/Group | Regular Eye
Number analyzed (Participants) | 42
normalized degree | -0.01 [-0.29 to 0.27]

ADVERSE EVENTS:
Arm/Group | Normal Eye | Large Regular Astigmatism | Large Irregular Astigmatism
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/34 | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor can require an extension of the embargo for 90 days. If the communication contains confidential information of the sponsor, the sponsor can require to replace this information by scientifically meaningful equivalent information.